CLINICAL TRIAL: NCT03284164
Title: An Open-Label Study to Investigate the Effect of Renal Impairment on the Pharmacokinectics of Tenofovir Exalidex
Brief Title: Evaluation of Effect of Renal Impairment on the PK of Tenofovir Exalidex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ContraVir Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: ContraVir (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRV-TXL-104
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-02

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Tenofovir exalidex (TXL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Subjects (Experimental): Healthy Subjects matched to RI subjects Tenofovir Exalidex (TXL)
  Interventions: Drug: Tenofovir Exalidex (TXL)
- Severe RI (Experimental): Severe Renal Impairment subjects Tenofovir Exalidex (TXL)
  Interventions: Drug: Tenofovir Exalidex (TXL)

INTERVENTIONS:
Drug: Tenofovir Exalidex (TXL) — Drug: Tenofovir Exalidex (TXL)
  Other Names: lipid conjugate TFV

SUMMARY:
This is a Phase 1 study to investigate the effects of Renal Impairment on the pharmacokinetics of Tenofovir exalidex

DETAILED DESCRIPTION:
This is a Phase 1 study to investigate the effects of Renal Impairment (mild, moderate and severe) on the pharmacokinetics of Tenofovir Exalidex

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years of age and over
* Capable of giving written informed consent
* Capable of completing study requirements

Exclusion Criteria:

* Positive result for HIV, HBV, or HCV
* History or medical condition which could impact patient safety
* Current or past abuse of alcohol or drugs
* Participation in another clinical trial within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacokinetics of TXL in subjects with RI compared to matching healthy volunteers | up to six days post dose
  Measuring Cmax : the peak plasma concentration

SECONDARY OUTCOMES:
Evaluation of the adverse events for TXL in RI subjects | up to six days post dose
  review of Adverse events
Evaluation of safety labs for TXL in RI subjects | up to six days post dose
  review of safety labs

CONTACTS AND LOCATIONS:
Overall Officials: John Sullivan-Bolyai, MD, MPH, Study Chair — ContraVir Pharmaceuticals
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided